CLINICAL TRIAL: NCT04124653
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, FIRST-IN-HUMAN STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE ASCENDING ORAL DOSES OF PF-06842874 ADMINISTERED AS AN IMMEDIATE-RELEASE OR MODIFIED-RELEASE FORMULATION TO HEALTHY ADULT PARTICIPANTS AND AN OPEN-LABEL ASSESSMENT OF THE RELATIVE BIOAVAILABILITY OF A MODIFIED-RELEASE FORMULATION OF PF-06842874
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PF-06842874 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C4041001
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Healthy Participants
Keywords: PF-06842874; first in human; cyclin-dependent kinase 4; cyclin-dependent kinase 6; CDK4/6; healthy participants; immediate release; modified release; relative bioavailability

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: participant- and investigator-blind, sponsor-open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06842874/Placebo (Experimental): Single dose administration of PF-06842874 or placebo
  Interventions: Drug: PF-06842874; Drug: Placebo
- Relative Bioavailability (Experimental): Determination of relative bioavailability of modified-release formulation relative to immediate-release formulation
  Interventions: Drug: Relative Bioavailability

INTERVENTIONS:
Drug: PF-06842874 — Single dose administration of PF-06842874
  Arms: PF-06842874/Placebo
Drug: Placebo — Single dose administration of placebo
  Arms: PF-06842874/Placebo
Drug: Relative Bioavailability — Relative bioavailability assessment of modified-release formulation
  Arms: Relative Bioavailability

SUMMARY:
This study will be the first time PF-06842874 is administered to humans. The purpose of Part A of the study is to investigate the safety, tolerability, and pharmacokinetics of PF-06842874 following administration of single oral doses as an immediate-release or modified-release formulation to healthy adult participants. Part B of this study will evaluate the relative bioavailability of a modified-release formulation of PF-06842874 for its potential use in future clinical studies. The effect of food on PF-06842874 pharmacokinetics may also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential and male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, and cardiac monitoring.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Any condition possibly affecting drug absorption.
* History of human immunodeficiency virus infection (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody.
* Participants with benign ethnic neutropenia or cyclic neutropenia.
* Other acute or chronic medical or psychiatric condition.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
* A positive urine drug test.
* Screening supine blood pressure (BP) ≥140 mmHg (systolic) or ≥90 mmHg (diastolic), following at least 5 minutes of supine rest.
* Baseline 12-lead standard electrocardiogram (ECG) that demonstrates clinically relevant abnormalities.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.25× upper limit of normal (ULN); total bilirubin level ≥1.5× ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN; hemoglobin ≤14 gm/dL (males) and ≤13 gm/dL (females); neutrophils <1500 cells/mm3.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of screening.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study medication
  Treatment-related AEs are any untoward medical occurrences attributed to study drug in a participant who received study drug.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 10 days after last dose of study medication
  The following parameters will be analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | 0, 1, 2, 3, 5, 8, 12, 24, and 48 hours post-dose
  The following parameters will be analyzed for examination of vital signs: systolic blood pressure, diastolic blood pressure, and pulse rate.
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | 0, 1, 2, 3, 5, 8, 12, 24, and 48 hours post-dose
  Measurements of heart rate, PR interval, QT interval, QTc intervals, and QRS complex
Abnormal rhythms as observed continuous cardiac monitoring | 0 to 8 hours post-dose
  Cardiac rhythms measured by continuous cardiac telemetry
Number of Participants With Clinically-Significant Change From Baseline in Physical Examination Findings | Baseline up to 10 days after last dose of study medication
  A complete physical examination includes, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A limited physical examination includes, at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant-reported symptoms.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-06842874 | 0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours post-dose
  Maximum observed plasma concentration for immediate-release and modified-release formulations of PF-06842874
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of PF-06842874 | 0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours post-dose
  Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration for immediate-release and modified-release formulations of PF-06842874
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-06842874 | 0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours post-dose
  Area under the plasma concentration versus time curve (AUC) from time zero to extrapolated infinite time (0-inf) for immediate-release and modified-release formulations of PF-06842874. It is obtained from AUC(0-t) plus AUC (t-inf).
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06842874 | 0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours post-dose
  Time to reach maximum observed plasma concentration for immediate-release and modified-release formulations of PF-06842874
Plasma Half-Life (t1/2) of PF-06842874 | 0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours post-dose
  Plasma half-life is the time measured for the plasma concentration to decrease by one half for immediate-release and modified-release formulations of PF-06842874.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Pfizer New Haven Clinical Research Unit, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4041001